CLINICAL TRIAL: NCT01911546
Title: A Prospective, Pilot Trial to Evaluate Safety and Tolerability of Everolimus for the Prevention of BK and CMV Viremia in HLA Sensitized Kidney Transplant Recipients
Brief Title: Role of Everolimus in Highly Sensitized Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph Kahwaji, MD, MPH (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Joseph Kahwaji, MD, MPH, former transplant nephrologist, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001AUS200T
Record Dates: First submitted 2013-03-04; First posted 2013-07-30 (Estimated); Results first posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-11

CONDITIONS: Highly-sensitized Kidney Transplant Recipients
MeSH Terms: interventions — Everolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- everolimus + low-dose tacrolimus (Experimental): Patients receiving everolimus will be on low dose tacrolimus.
  Interventions: Drug: everolimus + low-dose tacrolimus

INTERVENTIONS:
Drug: everolimus + low-dose tacrolimus — Patients are supplied everolimus (Zortress) + prograf
  Other Names: zortress + prograf

SUMMARY:
A growing number of patients on the kidney transplant waiting list are broadly human leukocyte antigen (HLA) sensitized (HS). These patients are unlikely to have a compatible donor. Therefore they wait longer and have increased morbidity and mortality. Desensitization with intravenous immune globulin (IVIG) and rituximab with alemtuzumab induction improves transplant rates and achieves good allograft outcomes. However, HS patients are at risk for viral infections after transplant. We have previously shown an increased incidence of BKV infections after desensitization with HS patients having higher peak viral loads. Cytomegalovirus (CMV) and polyomavirus BK (BKV) infections place HS renal transplant recipients at particular risk. Allograft rejection is associated with both CMV and BKV infection. This is of particular concern for HS patients as they are at an increased risk of rejection at baseline. Furthermore, the frequent development of leukopenia after transplantation often requires the CMV prophylactic agent to be discontinued along with lowering immunosuppression. This increases the risk of CMV infection and allograft rejection.

Everolimus was approved for rejection prophylaxis in combination with calcineurin inhibitors (CNI). CNI used in the study that led to drug's approval was cyclosporine. There are several trials nearing it's completion that utilize low dose tacrolimus instead. In 2012 Novartis published data from several trials showing superior outcomes using everolimus + low dose tacrolimus. This combination is currently approved in EU. It is also a combination that is standard of care (SOC) at our center for patients on everolimus.

This study aims to demonstrate that use of everolimus as part of a maintenance immunosuppression regimen may decrease viral infections without lowering overall immunosuppression thus improving allograft function and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Recipient of a deceased or living donor kidney allograft
2. Patients must have undergone desensitization with IVIG and rituximab with or without plasma exchange prior to transplant or be administered IVIG and rituximab peri-operatively.
3. Age 18 and over
4. Able to understand and provide informed consent

Exclusion Criteria:

Recipients of a dual simultaneous kidney/liver, kidney/heart, kidney/lung transplant 2. Pregnant or lactating females 3. Patients with a platelet count < 100,000/mm3 at time of randomization 4. Patients with an absolute neutrophil count < 1,500/mm3 or a white blood cell count of <3,000/mm3 at time of randomization 5. Patients who have an abnormal liver profile such as ALT, AST, Alkaline Phosphatase, or total bilirubin > 3 times the upper limit of normal (ULN) at time of randomization 6. Patients with severe total hypercholesterolemia (> 350 mg/dL; > 9 mmol/L) or total hypertriglyceridemia (> 500 mg/dL; > 5.6 mmol/L). Patients on lipid lowering treatment with controlled hyperlipidemia are acceptable.

7. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes 8. Patients being treated with drugs that are strong inducers or inhibitors of cytochrome P450 3A4 9. Patients with a clinically significant systemic infection within 30 days prior to transplant 9 10. Patients who have any surgical or medical condition, such as severe diarrhea, active peptic ulcer disease, or uncontrolled diabetes mellitus, which in the opinion of the investigator, might significantly alter the absorption, distribution, metabolism and/or excretion of study medication.

11. Patients with a history of coagulopathy or medical condition that would require long-term anticoagulation therapy after transplantation, unless the condition would permit a two week interruption in therapy before and after allograft biopsy. (Treatment with low dose aspirin is allowed.) 12. Women of childbearing potential who are either pregnant, lactating, planning to become pregnant during this trial, or with a positive serum or urine pregnancy test. Women of childbearing potential must be willing to agree to contraceptive practices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Highly HLA Sensitized Patients with End Stage Renal Disease Receiving Deceased Donor or Living Donor kidney transplant were enrolled.
Groups:
- Everolimus + Low-dose Tacrolimus: 20 patients received everolimus with low dose tacrolimus.
  Everolimus + low-dose tacrolimus: Patients are supplied everolimus (Zortress) + prograf
Period: Overall Study
Arm/Group | Everolimus + Low-dose Tacrolimus
Started | 20
Completed | 14
Not Completed | 6
Not completed — Lost to Follow-up | 1
Not completed — Everolimus was discontinued | 5

BASELINE CHARACTERISTICS:
Population: A total of 20 patients were enrolled in this clinical trial.
Units Other Than Participants: patients
Arm/Group | Everolimus + Low-dose Tacrolimus
Number analyzed (Participants) | 20
Number analyzed (patients) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.65 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 7
  More than one race | 7
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Cause of ESRD [Count of Participants; unit: Participants]
  Alport Syndrome | 1
  Congenital | 3
  FSGS | 2
  HTN | 3
  Lupus | 3
  PCKD | 2
  Post-Infectious Glomerulonephropathy | 1
  Unknown Etiology | 5

OUTCOME MEASURES:

1. Primary Outcome: The Number of Polyoma BK Viremia Patients
Description: Patients will be monitored at regular interval for the development of Polyomavirus Viremia.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus + Low-dose Tacrolimus
Number analyzed (Participants) | 20
Participants | 5

2. Primary Outcome: The Number of CMV Viremia
Description: The number of patients with CMV viremia
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus + Low-dose Tacrolimus
Number analyzed (Participants) | 20
Participants | 0

3. Primary Outcome: Incidence of Antibody Mediated Rejection (ABMR)
Description: Protocol biopsies were obtained at T0 and 6 months post transplant.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus + Low-dose Tacrolimus
Number analyzed (Participants) | 12
Participants | 2

4. Secondary Outcome: Incidence of Cell Mediated Rejection (CMR)
Description: Patients will be monitored for any episodes of CMR.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus + Low-dose Tacrolimus
Number analyzed (Participants) | 12
Participants | 2

ADVERSE EVENTS:
Time Frame: From transplant to 12 months post transplant.
Arm/Group | Everolimus + Low-dose Tacrolimus
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 9/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus + Low-dose Tacrolimus (N=20)
Edema (Renal and urinary disorders) | 1 (1) — Swelling was seen in patient one month post transplant
Urine Leak (Renal and urinary disorders) | 2 (2) — Urine leak occurred 2 weeks and 1 month post transplant
Antibody Mediated Rejection and Thrombotic Microangiopathy (Renal and urinary disorders) | 1 (1)
Antibody Mediated Rejection / FSGS /Small Bowel Obstruction/Dehydration (Renal and urinary disorders) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 1 (1)
Shortness of Breath and Atrial Fibrillation (Cardiac disorders) | 1 (1)
UTI (Renal and urinary disorders) | 1 (1)
Nocardia Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus + Low-dose Tacrolimus (N=20)
Headache (Nervous system disorders) | 5 (5)
Weakness (General disorders) | 2 (2)
Weight gain (Metabolism and nutrition disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 4 (4)
General pain (Nervous system disorders) | 8 (8)

LIMITATIONS AND CAVEATS:
There were a total of 20 patients enrolled into this clinical trial. Of the 20 patients, six patients were withdrawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No